CLINICAL TRIAL: NCT03093532
Title: A Hypertension Emergency Department Intervention Aimed at Decreasing Disparities
Acronym: AHEAD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Heather Prendergast, Professor, Vice Chair Clinical Affairs, Emergency Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2015-0323; R56HL126657 (NIH)
Record Dates: First submitted 2017-03-06; First posted 2017-03-28 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Hypertension
Keywords: emergency department; stage 2 hypertension; minorities
MeSH Terms: conditions — Hypertension; Emergencies | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research Assistants are blinded to study arm assignment of participant when assessing outcomes measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): The Usual Care group arm will received pre-printed discharge instructions and an outpatient referral. (This group represents standard of care.)
- ED SBIRT-HTN (Active Comparator): The ED SBIRT-HTN (The Emergency Department Screening Brief Intervention and Referral for Treatment) arm consists of a series of risk assessment tools (surveys, video, and noninvasive bedside assessments) designed to be efficient, patient-centered and educational for participants in an emergency department setting. Through the intervention, participants will learn more about hypertension management and complications associated with uncontrolled BP. Participants in the ED-SBIRT-HTN group will receive the following interventions:
  1) screening (risk assessment/stratification), 2) a limited bedside echocardiogram (looking for evidence of subclinical cardiac disease), and 3) a urine microalbumin test (marker of early cardiovascular disease).
  Interventions: Other: ED SBIRT-HTN
- E SBIRT-HTN + PACTH-c (Active Comparator): Participants randomized to the SBIRT-HTN +PACHT-c (Post-Acute Care Hypertension Transition Clinic) arm will receive all interventions of the ED SBIRT-HTN arm plus a 48-72 hour follow-up in the Post-Acute Care Hypertension Transition Clinic for repeat blood pressure assessment, review of screening assessments, and secured PCP appointment with a federally qualified health center within the study site's health system.
  Interventions: Other: ED SBIRT-HTN; Other: PACHT-c

INTERVENTIONS:
Other: ED SBIRT-HTN — Participants in the ED-SBIRT-HTN group will receive the following interventions:
  1) screening (risk assessment/stratification), 2) a limited bedside echocardiogram (looking for evidence of subclinical cardiac disease), and 3) a urine microalbumin test (marker of early cardiovascular disease).
  Other Names: Screening,Brief Intervention,Referral for Treatment HTN
  Arms: E SBIRT-HTN + PACTH-c; ED SBIRT-HTN
Other: PACHT-c — Participants randomized to the SBIRT-HTN +PACHT-c (Post-Acute Care Hypertension Transition Clinic) arm will receive all interventions of the ED SBIRT-HTN arm plus a 48-72 hour follow-up in the Post-Acute Care Hypertension Transition Clinic for repeat blood pressure assessment, review of screening assessments, and secured PCP appointment with a federally qualified health center within the study site's health system.
  Other Names: Post Acute Care Hypertension Transition Clinic
  Arms: E SBIRT-HTN + PACTH-c

SUMMARY:
Effective interventions that can address uncontrolled hypertension, particularly in underrepresented populations that use the emergency department (ED) for primary care, are critically needed. Uncontrolled hypertension (HTN) contributes significantly to cardiovascular morbidity and mortality and is more frequently encountered among patients presenting to the ED as compared to the primary care setting. EDs serve as the point of entry into the health care system for many high-risk patient populations, including minority and low-income patients. Based upon recent studies, the prevalence of uncontrolled/undiagnosed HTN in patients presenting to the ED is alarmingly high.

Thus emergency department engagement and early risk assessment/stratification is a feasible innovation to help close health disparity gaps in HTN.

This proposal involves a three-arm randomized controlled trial of 120 patients from the Emergency Department at University of Illinois Hospital with elevated blood pressure (BP) and no established primary care provider (PCP). The overarching goal is to improve follow-up rates and transition to PCP care at a federally qualified community health center (FQHC). The primary outcome will be blood pressure control. Secondary outcomes will be blood pressure improvement, treatment adherence, and hypertension knowledge. The central hypothesis of the proposal is that an ED-based screening, brief intervention, and referral for treatment program for HTN (SBIRT-HTN) using existing ED resources, coupled with a follow-up visit to an ED pharmacist-initiated Post-Acute Care Hypertension Transition Clinic (PACHT-c), can be impactful in a predominately underrepresented hypertensive population.

DETAILED DESCRIPTION:
Effective interventions to address uncontrolled hypertension (HTN), particularly in underrepresented populations that use the emergency department (ED) for primary care, are critically needed. Uncontrolled HTN, which contributes significantly to cardiovascular morbidity and mortality, is more frequently encountered among patients presenting to the ED. EDs serve as the point of entry into the health care system for many high-risk patient populations, particularly minority and low-income individuals. Our preliminary data from a largely minority patient population presenting to the ED shows significant rates of subclinical heart disease (diastolic dysfunction and left ventricular hypertrophy) in patients with elevated blood pressure (BP). These early echocardiogram changes are reversible with existing strategies for improving BP control.

The proposed project underscores that 1) The prevalence of uncontrolled/undiagnosed HTN among ED patients from underrepresented groups who do not have a primary care physician (PCP) is alarmingly high, and 2) ED engagement and early risk assessment/stratification with facilitated PCP follow-up is a novel and feasible innovation to help address health disparity gaps in HTN. The central hypothesis of the proposal is that an ED-based screening, brief intervention, and referral for treatment program for HTN (SBIRT-HTN) using existing ED resources, coupled with a follow-up visit to an ED pharmacist-initiated Post-Acute Care Hypertension Transition Clinic (PACHT-c), will improve BP control through patient empowerment, facilitating PCP follow-up rates, and consequently improving treatment compliance in a predominately underrepresented hypertensive population. This proposal is strengthened by the existing partnership between an academic urban ED and a Federally Qualified Health Center (FQHC) as a model for integrating secondary cardiovascular prevention in a population at high risk for complications due to uncontrolled/undiagnosed HTN. Moreover, this proposal is innovative as a prospective randomized controlled trial in a high-risk ED patient population with no established PCP and persistent elevated BPs.

Eligible patients are those with elevated BP and no established PCP (or no PCP contact in the past year) who present to the University of Illinois Hospital & Health Sciences System (UI Health) ED. The three arms are: 1) usual care (current practice of passive outpatient referral for follow-up care), 2) an ED-based SBIRT-HTN program (patient empowerment tool) using existing ED resources followed by assisted referral for usual care, and 3) the ED based SBIRT-HTN coupled with a 48-hour follow-up visit to an ED pharmacist-initiated Post-Acute Care Hypertension Transition Clinic (PACHT-c) followed by assisted referral for primary care.

The aims evaluate the effectiveness of the interventions (SBIRT-HTN & PACHTC-c) on uncontrolled BP at 6 months. The primary outcome will be BP improvement. Based on the demographics of the ED population at the study site (70% of the current UI Health ED population are ethnic minorities), the majority of participants will be underrepresented minorities (African-American and Hispanic/Latino) and low-income individuals. The investigators propose the following specific aims and hypotheses:

Aim 1: Evaluate the effectiveness of an ED-initiated SBIRT-HTN program on BP control at 6 months post intervention compared to usual care.

H1: Early identification and initiation of a risk stratification algorithm that involves non-invasive assessment (limited echocardiogram) for early subclinical cardiovascular disease (combined with patient education regarding HTN & cardiovascular complications (patient empowerment) at the point-of contact in the ED (arm 2) will result in greater BP control at 6 months compared to the usual care group (arm 1).

Aim 2: Evaluate the impact of the PACHT-c component with the ED-based SBIRT-HTN program on BP control at 6 months post intervention compared to usual care and ED-SBIRT-HTN alone.

H2: The PACHT-c component (arm 3) will result in greater BP control compared to those randomized to usual care (arm 1) or ED-based SBIRT-HTN alone (arm 2).

ELIGIBILITY:
Inclusion Criteria:

* Stage 2 Hypertension- Elevated BP of ≥160/100 at time of discharge from ED
* Verbal fluency in English or Spanish
* Age 30 to 64 years

Exclusion Criteria:

* Unable to verbalize comprehension of study or impaired decision making (e.g., dementia)
* History of heart failure, myocardial infarction, or stroke
* Lives outside Chicago communities
* Plans to move from Chicago area within the next year
* Pregnant or trying to get pregnant

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Control (BP < 140/90 mmHg) at 6 Months | 6 months
  In order to be eligible for the study, patients must have uncontrolled BP. At 6 months, we will determine if patients have controlled their BP, as evidenced by BP < 140/90 mmHg.
  BP measurements will be recorded on seated participants after at least five minutes in a quiet room. ED-pharmacists and trained research assistants will perform BP, measurements using digital BP meters using standardized procedures.

SECONDARY OUTCOMES:
Change from Baseline Blood Pressure (Systolic/Diastolic mm Hg) at 6 Months | 0, 6 months
  Blood pressure will be collected at two time points (baseline and 6 months). BP measurements will be recorded on seated participants after at least five minutes in a quiet room. ED-pharmacists and trained research assistants will perform BP, measurements using digital BP meters using standardized procedures.
Change in Hypertension Knowledge at 6 Months (Hypertension Knowledge Survey) | 0, 6 months
  The hypertension knowledge survey is a 10-item, validated tool developed to assess hypertension knowledge in low literacy patient populations. The scale assesses respondents' knowledge in defining hypertension, lifestyle, and behaviors that may affect BP levels, and the long-term consequences of HTN. The survey has been validated in an urban population that included a high proportion of black and Latino patients. Scores are categorized into tertiles that indicate low (≤7), medium (8), or high (9-10) levels of HTN knowledge.
Change in Treatment Adherence at 6 Months (Modified Morisky Scale) | 0, 6 months
  The modified Morisky scale is a validated 4-item instrument to assess self-reported patient adherence related to antihypertensive medication. The modified Morisky scale provides a total score with a range of 0 to 4, with higher scores indicating lower adherence to medication. The scores of the modified Morisky scale can be classified as low compliers (3-4), medium compliers (1-2) and high compliers (0) based on its criterion validity with BP control.

IPD SHARING:
Plan to Share IPD: No